CLINICAL TRIAL: NCT01992705
Title: Neoadjuvant FOLFIRINOX and Stereotactic Body Radiotherapy (SBRT) Followed by Definitive Surgery for Patients With Borderline Resectable Pancreatic Adenocarcinoma: A Single-Arm Pilot Study
Brief Title: Borderline Pancreas Study: FOLFIRINOX +SBRT
Acronym: GCC 1324
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00055716
Record Dates: First submitted 2013-09-27; First posted 2013-11-25 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Resectable Pancreatic Cancer
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy+SBRT prior to surgery if applicable (Other): FOLFIRINOX Drugs:
  * Calcium Folinate (Folinic Acid) 400 mg IV on Day 1 of each cycle (21d/cycle for a total of 4 cycles.
  Stereotactic Body Radiotherapy (SBRT):
  30 Gy in 5 fractions given to radiographically defined pancreatic mass alone
  Interventions: Other: Chemotherapy(FOLFIRINOX) + SBRT prior to surgery if applicable; Drug: -Oxaliplatin 85 mg/m2 IV on Day 1; Drug: -Irinotecan 180 mg/m2 IV on Day 1; Drug: -5-FU (Fluorouracil) 2,400 mg/m2 IV over 46-48 hours

INTERVENTIONS:
Other: Chemotherapy(FOLFIRINOX) + SBRT prior to surgery if applicable — Patients will receive chemotherapy (21d/cycle for a total of 4 cycles) plus SBRT before screening for surgical resection of the pancreas.
Drug: -Oxaliplatin 85 mg/m2 IV on Day 1 — Oxaliplatin 85 mg/m2 IV on Day 1 of each cycle (21d/cycle for a total of 4 cycles).
Drug: -Irinotecan 180 mg/m2 IV on Day 1 — Irinotecan 180 mg/m2 IV on Day 1 of each cycle (21d/cycle for a total of 4 cycles).
Drug: -5-FU (Fluorouracil) 2,400 mg/m2 IV over 46-48 hours — 5-FU (Fluorouracil) 2,400 mg/m2 IV over 46-48 hours of each cycle (21d/cycle for a total of 4 cycles.

SUMMARY:
Primary Objective: To determine the rate of downstaging to resectability in patients with borderline resectable pancreatic cancer receiving FOLFIRINOX and SBRT as preoperative therapy.

Secondary Objective(s):

1. To assess the disease-free-survival, overall survival, time to recurrence and site of recurrence in patients with borderline resectable pancreatic cancer receiving preoperative FOLFIRINOX followed by SBRT
2. To investigate the safety and tolerability of FOLFIRINOX and SBRT in patients with resectable pancreatic cancer
3. To determine the radiologic and pathological response associated with preoperative SBRT and FOLFIRINOX therapy
4. To assess quality of life through and after treatment using the FACT-Hep questionnaire

DETAILED DESCRIPTION:
The study investigators hypothesize that neoadjuvant FOLFIRINOX can be safely and efficaciously delivered using a sequential regimen with SBRT as an alternative to standard neoadjuvant chemoradiotherapy. Standard of care neoadjuvant treatment typically requires about six weeks of treatment with sub-systemic dosing of chemotherapy. The feasibility of the sequential delivery of the FOLFIRINOX followed by SBRT will be evaluated by capturing the prevalence of grade 3 toxicity and the treatment delay rate.

In our study, SBRT is planned sequentially to follow cycle 4 of chemotherapy treatment, provided toxicity has resolved to grade 2 or less. Thus, allowing for resolution of chemotherapy toxicity prior to initiation of radiation therapy. This interval and the fact that there is no concurrent delivery of chemo-RT, based on previously discussed experiences, including approaches where SBRT safely follows other intense chemotherapy regimens (see Polistina et al and Chuong [35,36]) makes this study feasible without establishing toxicity profile.

The proposed regimen of 4 cycles of FOLFIRINOX followed by 30 Gy/5 fractions using SBRT will be safely tolerated and will improve resectability rates in borderline resectable PDAC patients. In addition, this regimen will not compromise the ability to achieve a successful Whipple resection.

This regimen will improve the local control rate and overall disease free survival in this patient population. The investigators further hypothesize that early administration of FOLFIRNOX will provide optimal systemic therapy to control clinically occult micrometastases.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years at diagnosis.
* Biopsy proven pancreatic adenocarcinoma.
* Borderline resectable per NCCN criteria (No distant metastases, venous involvement of the portal vein/SMV, demonstrating tumor abutment and narrowing of the lumen, encasement of the portal vein/SMV without encasement of the nearby arteries, or short-segment venous occlusion resulting from either tumor thrombus or encasement but with suitable vessel proximal or distal to this area of vessel involvement, allowing for safe resection and reconstruction; gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery, without extension to the celiac axis; tumor abutment of the SMA not to exceed 180 degrees of the circumference of the vessel wall.).
* Radiologically measurable or clinically evaluable disease.
* Pancreas protocol CT and/or MRI if required for further clarification of disease tissue planes within 4 weeks of registration.
* ECOG PS of 0-2.
* Able to get a Whipple resection per surgeon assessment performed within 4 weeks of registration.
* The following laboratory values obtained ≤ 28 days prior to registration:
* Absolute neutrophil count (ANC) ≥ 1,500/mm3.
* Platelet count ≥ 100,000/mm3.
* Hemoglobin > 8.0 g/dL.
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN).
* SGOT (AST) ≤ 2 x ULN.
* SGPT (ALT) ≤ 2 x ULN.
* Creatinine ≤ 1.5 x ULN.
* CA 19-9 level (to establish baseline).
* A negative pregnancy test within 7 days prior to registration for women of childbearing potential. In addition, male and female participants must commit to adequate contraception while on study.
* Able to provide written informed consent.
* Willing to return for all required study assessments.
* Neurological assessment for pre-existing peripheral neuropathy.
* Documentation of pre-existing hearing deficits.

Exclusion Criteria:

* Any pancreatic adenocarcinoma that does not meet criteria for borderline resectable disease.
* Prior history of abdominal radiation therapy.
* History of autoimmune disease such as scleroderma, lupus, and inflammatory bowel disease.
* Patients with tumor-caused symptomatic bowel obstruction.
* Chemotherapy (including hormonal therapy) within the past 5 years from date of registration.
* Other invasive malignancies within the past 5 years from date of registration.
* Pregnant or nursing women or women of childbearing age that are unwilling to employ adequate contraception.
* Other co-morbid conditions which, based on the judgment of the physicians obtaining informed consent, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-03; Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Rate of downstaging to resectability in patients with borderline resectable pancreatic cancer receiving FOLFIRINOX and SBRT as preoperative therapy. | Participants will be followed from randomization up to 120 months or death (from any cause) whichever comes first.
  To determine the rate of downstaging to resectability in patients with borderline resectable pancreatic cancer receiving FOLFIRINOX and SBRT as preoperative therapy (AGGC 6th edition).

SECONDARY OUTCOMES:
Survival status (disease-free-survival vs. overall survival) time to recurrence and site of recurrence in patients with borderline resectable pancreatic cancer receiving preoperative FOLFIRINOX followed by SBRT | Participants will be followed from randomization up to 120 months or death (from any cause) whichever comes first.
  To assess the disease-free-survival, overall survival, time to recurrence and site of recurrence in patients with borderline resectable pancreatic cancer receiving preoperative FOLFIRINOX followed by SBRT (RECIST)

OTHER OUTCOMES:
Number of adverse events/toxicites reported during and following treatment of FOLFIRINOX and SBRT in patients with resectable pancreatic cancer | Participants will be followed from randomization up to 120 months or death (from any cause) whichever comes first.
  Number of toxicities participants reported by participants during and following treatment with FOLFIRINOX and SBRT in patients with resectable pancreatic cancer (NIH CTCAE v.4).
Radiologic and pathological response associated with preoperative SBRT and FOLFIRINOX therapy | Participants will be followed from randomization up to 120 months or death (from any cause) whichever comes first.
  To determine the radiologic and pathological response associated with preoperative SBRT and FOLFIRINOX therapy (review of radiology and pathology reports).
Quality of life through and after treatment | Participants will be followed from randomization up to 120 months or death (from any cause) whichever comes first.
  To assess quality of life through and after treatment using the FACT-Hep questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shahed Badiyan, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States